CLINICAL TRIAL: NCT03869567
Title: Cone Beam Computed Tomography Following Thrombectomy : Identification of Hemorrhage and Distinction From Contrast Accumulation Due to Blood-Brain Barrier Disruption
Brief Title: Cone Beam Computed Tomography Following Thrombectomy
Acronym: Hemathromb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0027
Record Dates: First submitted 2019-02-21; First posted 2019-03-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Hemorrhage
Keywords: thrombectomy; flat panel Computed tomography; cone beam computed tomography; hemorrhage; stroke; dual energy computed tomography
MeSH Terms: conditions — Stroke; Hemorrhage | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cone beam CT (Experimental): A cone beam CT wll be performed just after thrombectomy on patients with acute ischemic stroke
  Interventions: Device: cone beam CT

INTERVENTIONS:
Device: cone beam CT — Just after thrombectomy, a cone beam CT will be done, while patient is on angiography table, in order to determine if hemorrhage image is due to contrast accumulation or blood-brain barrier disruption.

SUMMARY:
Cerebral haemorrhages following reperfusion treatments involve not only rupture of the blood-brain barrier, but also direct damage to vessels related to the equipment used and secondary toxicity to thrombolytics. The rupture of the blood-brain barrier which results from ischemia / reperfusion is responsible for stagnation of the contrast product on the exams performed after thrombectomy. It is difficult to distinguish hyperdensities related to the stagnation of contrast product and Hemorrhage on a conventional scanner. The reference imaging is the double energy scanner performed at the thrombectomy outlet. But no study directly compared the results of the flat panel with the cone beam CT performed in immediate post-thrombectomy. The investigators propose a direct comparison of the cone beam CT with the dual energy CT performed at the exit of thrombectomy.

DETAILED DESCRIPTION:
Until December 2014, intravenous thrombolysis was the only reperfusion therapy proven to be effective within 4 hours of a cerebral infarction and several studies showed a clear functional benefit of thrombectomy in combination with thrombolysis in the first six hours of proximal arterial occlusion. Cerebral haemorrhages following reperfusion treatments involve not only rupture of the blood-brain barrier, but also direct damage to vessels related to the equipment used and secondary toxicity to thrombolytics. The rupture of the blood-brain barrier which results from ischemia / reperfusion is responsible for stagnation of the contrast product on the exams performed after thrombectomy, but it is difficult to distinguish hyperdensities related to the stagnation of contrast product and Hemorrhage on a conventional scanner. Several techniques are available to evaluate the hyperdensities post endovascular cerebral reperfusion including: the dual energy ct, the flat panel CT performed in the angiography room and the conventional scanner. The Cone beam CT is a relevant exam because it is performed in the angiography room and does not require transporting the patient who can be agitated or intubated until the scanner. The reference imaging is the double energy scanner performed at the thrombectomy outlet. Some studies have shown an excellent negative predictive value of the flat panel CT to eliminate haemorrhage in post-thrombectomy but no study directly compared the results of the flat panel with the CT performed in immediate post-thrombectomy and even less with the double energy scanner, it is therefore difficult to assert the sensitivity and exact specificity of this exam to detect and distinguish haemorrhage from contrast stagnation. The investigators propose a direct comparison of the cone beam CT with the dual energy CT performed at the exit of thrombectomy.

Method: consecutive patients presenting acute ischemic stroke candidates to thrombectomy will be enrolled in one hospital center. A cone beam Ct will be performed at the end of the procedure as well as a dual energy CT and finally a CT 24 h after the thrombectomy. Predictive factors of hemorrhage transformation such blood barrier disruption will be studied secondarily.

ELIGIBILITY:
Inclusion Criteria:

* all patients with cerebral thrombectomy
* Adults
* Patients able to express consent
* Signed written informed consent form
* Covered by national health insurance

Exclusion Criteria:

* minors
* pregnancy or beast feeding
* patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)
* obstruction to participate
* non covered by national health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage presence | up to two days
  hemorrhage presence or not is determined with cone beam and scanner images

SECONDARY OUTCOMES:
Number of patients with hemorrhagic transformation | 24 hours from symptom onset
  Any type of parenchyma hemorrhage according to ECASS II criteria (European Cooperative Acute Stroke Study 2). Scores are HI1, HI2, PH1 or PH2. HI1 = small petechia around stroke area. HI2 = confluent petechia in the stroke area. PH1 = Hematoma with less than 30% stroke weight. PH2 = Hematoma with more than 30% stroke weight.
Health deterioration | 24 hours from symptom onset
  Any deterioration in NIHSS score (NIHSS : National Institute of Heath Stroke ) or death combined with intracerebral hemorrhage. Scale of NIHSS score : 1 to 42. Minimum score : 1. Maximum score : 42. 1-4 : minor stroke. 5-15 : mild stroke. 15-20 : acute stroke. More than 20 : major stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Chivot, Dr, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No